CLINICAL TRIAL: NCT00465556
Title: Domestic Violence Enhanced Home Visitation Program - DOVE
Brief Title: Domestic Violence Enhanced Home Visitation Program (DOVE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Phyllis Sharps, Professor, Associate Dean, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NR009093; 1R01NR009093-01A2 (NIH)
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Domestic Violence
MeSH Terms: interventions — Poliovirus Vaccine, Inactivated; Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Dove Intervention
  Interventions: Behavioral: Public Health Nurse Home Visit
- 2 (Active Comparator): Intimate Partner Violence (IPV) Protocol
  Interventions: Behavioral: Intimate Partner Violence (IPV) Protocol

INTERVENTIONS:
Behavioral: Public Health Nurse Home Visit — The perinatal public health nurse home visit intervention also includes a trifold brochure, printed on 8X10 inch paper, with 6 panels, that can be read with the woman in an interactive manner so that the woman is encouraged to describe her experiences and choose her options as they proceed. Participants will receive three prenatal and three postpartum sessions. The first prenatal sessions will be given during the first (enrollment), second, and third trimesters, with at least three weeks between sessions. Women entering the study after the first trimester will receive the initial session at enrollment, with two subsequent sessions spread out over the remainder of the scheduled prenatal home visitation program sessions.
  Arms: 1
Behavioral: Intimate Partner Violence (IPV) Protocol — The current protocol in use by the participating health departments when a women screens positive for intimate partner violence (IPV), current or history within the last year.
  Arms: 2

SUMMARY:
DOVE Home Visit Program is a brochure based intervention delivery by public health nurses which aims to prevent and reduce intimate partner violence against pregnant and postpartum women and their infants.

The purpose of the study is to test the effect of home visits on reducing domestic violence and improving the lives of pregnant women and their children.

DETAILED DESCRIPTION:
Outcomes will provide intervention efficacy data about a public health nurse home visit intervention aimed at reducing and preventing intimate partner violence and children's exposure to IVP as well as prospective information about patterns of intimate partner violence.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 31 weeks or less gestation, over age 18, with a history of intimate partner violence within the past 2 years, and who are willing to participate in the home visit program

Exclusion Criteria:

Age 17 or less. History of partner violence beyond 2 years. Not participating in home visit program. Does not speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2006-02; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Reducing children's exposure to Intimate Partner Violence | Baseline (entry into the study), birth of the infant, and 3, 6, 12 and 24 months after the infant's birth.
Patterns of Intimate Partner Violence | Baseline (entry into the study), birth of the infant, and 3, 6, 12 and 24 months after the infant's birth.
Reducing Intimate Partner Violence | Baseline (entry into the study), birth of the infant, and 3, 6, 12 and 24 months after the infant's birth.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Sharps, PhD, RN, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Baltimore City Health Department, Baltimore, Maryland
  - Missouri Department of Health and Senior Services; Missouri Community Based Home Visiting Program and Lutheran and Family Children's Services in Columbia and Springfield, Columbia, Missouri

REFERENCES:
- [Derived] Kalra N, Hooker L, Reisenhofer S, Di Tanna GL, Garcia-Moreno C. Training healthcare providers to respond to intimate partner violence against women. Cochrane Database Syst Rev. 2021 May 31;5(5):CD012423. doi: 10.1002/14651858.CD012423.pub2. PMID 34057734
- [Derived] Sharps PW, Bullock LF, Campbell JC, Alhusen JL, Ghazarian SR, Bhandari SS, Schminkey DL. Domestic Violence Enhanced Perinatal Home Visits: The DOVE Randomized Clinical Trial. J Womens Health (Larchmt). 2016 Nov;25(11):1129-1138. doi: 10.1089/jwh.2015.5547. Epub 2016 May 20. PMID 27206047
- [Derived] Sharps P, Alhusen JL, Bullock L, Bhandari S, Ghazarian S, Udo IE, Campbell J. Engaging and retaining abused women in perinatal home visitation programs. Pediatrics. 2013 Nov;132 Suppl 2(Suppl 2):S134-9. doi: 10.1542/peds.2013-1021L. PMID 24187115